CLINICAL TRIAL: NCT00241124
Title: A Randomized, Double Blind, Double Dummy, Parallel Group, Active-Controlled Study To Evaluate The Effectiveness Of Morning Versus Evening Doses Of 320 Mg Valsartan Versus 40 Mg Lisinopril On The 24 Hour Blood Pressure Profile In Patients With Hypertension And Non-Insulin Dependent Diabetes
Brief Title: Comparison Of Morning And Evening Dosing Of Valsartan And Lisinopril In Patients With Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAL489A2420
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension
Keywords: hypertension; valsartan; morning/evening dosing; lisinopril
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Lisinopril

INTERVENTIONS:
Drug: valsartan
Drug: lisinopril

SUMMARY:
A study comparing the antihypertensives Valsartan and Lisinporil when doses are in the morning and comparing a morning dose of Valsartan with an evening dose.

ELIGIBILITY:
Inclusion Criteria:

- Hypertension defined by a MSSBP >=150 mmHg (untreated patients) or patients on current anti-hypertensive treatment who remain uncontrolled (i.e. MSSBP >140 mmHg)

* Randomisation mean 24h blood pressure above 130/80 mmHg
* In addition the patients must fulfill, at least, one of the following criteria:

Controlled type II Diabetes mellitus Hypercholesteremia, currently treated with lipid-lowering drugs Metabolic syndrome MI, CABG or PTCA more than one year ago Stroke or transient ischemic cerebral attack more than one year ago Documented history of peripheral vascular disease, increased IMT, or carotid plaques Documented history of LVH Elderly >65 years

Exclusion Criteria:

* - MSSBP >=180 mmHg and/or MSDBP >= 110 mmHg at any time from Visit 1 to Visit 3
* Inability to discontinue all prior anti-hypertensive medications safely for a period of three weeks
* Mandatory indication for any concomitant medication for coronary artery disease or any other disease that is not allowed during this study.

Other protocol-defined exclusion criteria may apply.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1099 (Actual)
Dates: Start 2004-04; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Average 24 hour blood pressure less than 130/80 mmHg after 26 weeks
Change from baseline in systolic 24 hour blood pressure after 12 weeks

SECONDARY OUTCOMES:
Change from baseline manual blood pressure and pulse pressure after 26 weeks
Change from baseline markers of endothelial function, fibrosis, and other blood measurements of hypertension after 12 and 26 weeks
Changes in ambulatory blood pressure measurements at various timepoints up to 26 weeks
Change from baseline heart size after 26 weeks
Adverse events, serious adverse events, laboratory values, physical examinations, vital signs for up to 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Investigative Centers, Germany

REFERENCES:
- [Derived] Zappe DH, Crikelair N, Kandra A, Palatini P. Time of administration important? Morning versus evening dosing of valsartan. J Hypertens. 2015 Feb;33(2):385-92. doi: 10.1097/HJH.0000000000000397. PMID 25259546